CLINICAL TRIAL: NCT04719052
Title: Mediterranean Enriched Diet for Tackling Youth Obesity
Acronym: MED4Youth
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fundació Eurecat (Other)
Collaborators: University of Parma (Other); University of Coimbra (Other); Hospital Universitari Sant Joan de Reus (Other)
Responsible Party: Principal Investigator, Antoni Caimari, Director of Eurecat's Biotechnology Area, Principal Investigator, Fundació Eurecat
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1
Record Dates: First submitted 2021-01-14; First posted 2021-01-22 (Actual); Last update posted 2024-10-30 (Actual); Status verified 2024-10

CONDITIONS: Obesity, Adolescent; Lifestyle, Healthy; Diet, Healthy; Cardiovascular Risk Factor
Keywords: Youth Obesity; Mediterranean diet; Interventional study; Healthy lifestyles; Educational approach
MeSH Terms: conditions — Pediatric Obesity | interventions — Diet; Diet, Mediterranean; Diet, Fat-Restricted

STUDY DESIGN:
Intervention Model Description: A multicentre, blind, single-randomized, parallel, clinical trial
Who Masked: Investigator
Masking Description: Due to the nature of the study, the participants cannot be blinded to the intervention, although the investigators who will perform the sample and data analysis will be blinded.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mediterranean diet group (Experimental): 1) The MD will be based on high consumption of unsaturated fat from vegetable sources (virgin olive oil and nuts) and minimally processed plant foods (vegetables, fruits, nuts, whole grains and legumes), low consumption of meat (especially red and processed meats) and sweets, and moderate consumption of fish and dairy products (mainly yoghurt and cheese). Accordingly, this diet will provide a high amount of mono and polyunsaturated fatty acids, fibre and phenolic compounds.
  Adolescents in the MD group will replace the intake of conventional breads by sourdough bread consumption (2 servings of 50-60 g daily) and incorporate into their diet chickpeas (2 servings of 150 g/week chickpeas, minimum one of them in hummus format), and they will consume at least another serving of legumes which can be chickpeas or another legume), pomegranate juice (4 servings of 200ml/week) and mixed nuts (4 servings of 30 g/week).
  Interventions: Other: Diet and behavioural intervention
- Low-fat diet group (Active Comparator): 2) The low-fat diet (control diet) will be based on low consumption of fats. A low-fat diet is the most used diet for obesity treatment in adolescents. This group will not receive any additional specific food by researchers. This diet will be based on the diet proposed as low-fat diet in the PREDIMED study
  Interventions: Other: Diet and behavioural intervention

INTERVENTIONS:
Other: Diet and behavioural intervention — Intervention will receive a specific diet designed following the characteristics of Mediterranean Diet
  Other Names: MEDITERRANEAN DIET
  Arms: Mediterranean diet group
Other: Diet and behavioural intervention — Control group will receive a specific diet designed following the characteristics of Low fat Diet.
  Other Names: LOW-FAT DIET
  Arms: Low-fat diet group

SUMMARY:
The prevalence of obesity is one of the main public health problems worldwide, reaching 18% among young people between 5 and 19 years of age in 2016. One possibility of effective treatment can be the Mediterranean diet (MD). Therefore, it is proposed to carry out a nutritional intervention based on this diet to more effectively reduce obesity in adolescents. The main purpose of this multicentre study is to assess whether an energy-restricted Mediterranean-style diet (MD) intervention including healthy products from the Mediterranean basin (mixed nuts, pomegranate and hummus) and sourdough bread is more effective against obesity and associated CVD risk factors than a conventional low-fat diet carrying out a multicentre nutritional and clinical intervention study specifically targeting obese/overweight adolescents (13-17y) from different Mediterranean countries; all combined with an educational web-application designed to encourage healthy behaviours.

It is a multicenter, randomized, controlled intervention study conducted with adolescents with obesity/overweight ≥90 percentile who do not suffer from any chronic disease. 240 subjects will be recruited from three Mediterranean countries: Italy (Parma), Portugal (Coimbra) and Spain (Reus), specifically 80 participants per country, 40 adolescents as an intervention group and 40 as a control group, in Reus. The intervention study is scheduled to begin in January 2021.

The intervention group will receive a diet based on the characteristics of MD, and will be reinforced with satisfying and healthy Mediterranean foods such as sourdough bread (2 servings of 50-60g / day), squeezed pomegranate (4 servings of 200ml / week), hummus/chickpeas (2 portions of chickpeas of 150-200g / week, one in hummus format) and mixed nuts (4 servings of 30g / week); and the control group will receive a recommended diet based on the consumption of low-fat foods. A caloric restriction of 20% of the total energy requirements will be applied to both groups in adolescents with BMI ≥95 percentile (obesity) and a caloric restriction <20% of the total energy requirements will be applied in adolescents with BMI ≥90 to <95th percentile according to overweight (gender/age / physical activity). The diet will be applied for 4 months in both groups. Adolescents from both groups will be given a motivational interview and will be provided with an educational website that will be used during the intervention, through which they will learn.

DETAILED DESCRIPTION:
The principal outcome is BMI z-score, a standardized measure of BMI based on the specific age and gender norms. The effectiveness of the intervention will be evaluated by comparing the BMI z-score between the control (low-fat diet) and intervention (MD) groups.

The secondary outcomes are: Adherence to the DM, KidMed questionnaire; Level of physical activity, PAQ-A questionnaire; Habit/food intake: 3-day dietary record, Helena study food frequency questionnaire, Knowledge about food and nutrition, a questionnaire from Helena's study; Quality of life, kid screen-27 Index; Sociodemographic data of the parents; Anthropometric data: weight, height, BMI, body composition, waist circumference, waist-hip ratio; Clinical variables: blood pressure, Biochemical variables and omic determinations: in urine, blood and feces.

In total, the adolescents will receive 5 visits:

* 1 pre-selection visit (to check inclusion / exclusion criteria in the study) (V0)
* 1 inclusion visit (V1) in which stool, urine, and blood samples will be collected, anthropometric measurements (such as weight and waist circumference) and blood pressure will be taken, and questionnaires and records will be answered dietary.
* 1 follow-up visit (V2), at 2 months, in which anthropometric and blood pressure measurements will be taken and questionnaires and dietary records will be answered.
* 1 final visit (V3), at 4 months, in which stool, urine, and blood samples will be collected, anthropometric and blood pressure measurements will be made, and questionnaires and dietary records will be answered.
* 1 post-intervention follow-up visit (V4), 4 months after the end of the intervention, in which anthropometric and blood pressure measurements will be taken and questionnaires and dietary records will be answered.

ELIGIBILITY:
Inclusion Criteria:

* boys and girls aged 13-17 years
* having obesity, defined as an age- and sex-specific BMI in the 95th percentile or greater (1), or great overweight (age- and sex-specific BMI in the ≥90th to <95th percentile),
* having informed consent (sign by both, one parent and the adolescent),
* and to have a mobile phone with internet access.

Exclusion Criteria:

* having diabetes and other metabolic, endocrine and chronic disorders;
* intake of antibiotics, drug, probiotics or nutritional supplements in the last month;
* prescribed medicine to control hypertension, inflammation or dyslipidemia,
* following a prescribed diet for any reason, including weight loss, in the last 3 months;
* following a religion-restricted diet;
* and having allergies or food intolerances in: nuts, pomegranate, bread and/or chickpeas.

Ages: 13 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 240 (Actual)
Dates: Start 2021-05-25 (Actual); Primary Completion 2023-10-09 (Actual); Study Completion 2023-11-28 (Actual)

PRIMARY OUTCOMES:
Change from baseline BMI z-score at 4 months and 8 months | "4 months" and "4 months after study cessation"
  The principal outcome is BMI z-score, a standardized measure of BMI based on the specific age and gender norms. The effectiveness of the intervention will be evaluated by comparing the BMI z-score between the control (low-fat diet) and intervention (MD) groups.

SECONDARY OUTCOMES:
Change from baseline Adherence to the Mediterranean Diet at 4 and 8 months | "4 months" and "4 months after study cessation"
  Change of Adherence to the Mediterranean Diet using KIDMED test by comparing control between the intervention group
  Scores:
  =<3 points: Very low-quality diet 4 to 7 points: Need to improve the eating pattern to fit the model Mediterranean.
  =>8 points: Optimal Mediterranean diet
Change from baseline Level of physical activity at 4 and 8 months | "4 months" and "4 months after study cessation"
  Change of Physical Activity using the Physical Activity Questionnaire test by comparing control between the intervention group A score 1 indicates low physical activity whereas a score of 5 indicates high physical activity
Change from baseline Habit/food intake at 4 and 8 months | "4 months" and "4 months after study cessation"
  Change of Habit/food intake using 3-day dietary record, Helena study food frequency questionnaire by comparing control between intervention group
Change from baseline Knowledge about food and nutrition intake at 4 and 8 months | "4 months" and "4 months after study cessation"
  Change of Knowledge about food and nutrition intake using Helena's study knowledge questionnaire by comparing control between intervention group
Change from baseline Life quality at 4 and 8 months | "4 months" and "4 months after study cessation"
  Change of life quality using kidscreen-27 Index by comparing control between intervention group
Sociodemographic data of the parents one time frame | 1 time frame
  Sociodemographic data of the parents will be assessed at baseline of study using Healthy Behaviour in School Age Children. Sociodemographic data will be divided by low, medium or high socioeconomic level.
Change from baseline BMI data at 4 and 8 months | "4 months" and "4 months after study cessation"
  BMI will be assessed by weight (kg) / height (m2), and using Centers for Disease Control and Prevention (CDC) BMI percentiles and will be compared between control and intervention group.
Change from baseline waist circumference data at 4 and 8 months | "4 months" and "4 months after study cessation"
  Waist circumference (cm) will be evaluated and will be compared between control and intervention group.
Change from baseline Waist-hip ratio data at 4 and 8 months | "4 months" and "4 months after study cessation"
  Waist-hip ratio will be evaluated by waist and hip circumference and will be compared between control and intervention group.
Change of Gut-derived metabolites (LPS, SCFAs, lactate, bile acids) | 4 months
  Gut-derived metabolites of both groups will be evaluated by Faeces and/or plasma using NMR /GC-MS
Change of biomarkers of oxidative stress (8-OHdG, F2-isoprostanes) | 4 months
  Biomarkers of oxidative stres of both groups will be evaluated by urine using ELISA
Change of biomarkers of inflammation (IL-6, CRP, TNFα, MCP1, IL-8) | 4 months
  Biomarkers of inflammation of both groups will be evaluated by plasma using Magnetic bead-based multiplex assays Homeostatic Model Assessment for insulin resistance
Change of biomarkers of adipose tissue function (adiponectin, leptin, resistin) | 4 months
  Biomarkers of adipose tissue function of both groups will be evaluated by plasma using Magnetic bead-based multiplex assays Homeostatic Model Assessment for insulin resistance
Change of Biomarkers of insulin resistance | 4 months
  Biomarkers of insulin resistance of both groups will be evaluated by plasma using Magnetic bead-based multiplex assays Homeostatic Model Assessment for insulin resistance
Change of biomarkers of cardiovascular risk (TMAO) | 4 months
  Biomarkers of cardiovascular risk of both groups will be evaluated by plasma and urine using UHPLC MS
Change of circulating levels of glucose and blood lipid profile | 4 months
  Circulating levels of glucose and blood lipid profile of both groups will be evaluated using Enzymatic assays
Change of Food Intake biomarkers | 4 months
  Food Intake biomarkers of both groups will be evaluated by urine using Metabolomics (UHPLC MS)
Change of Advanced glycation end products (AGEs) related analyses | 4 months
  Advanced glycation end products will be assessed by plasma or erythrocytes using ELISA / enzymatic assays

CONTACTS AND LOCATIONS:
Overall Officials: Antoni Caimari, PhD, Principal Investigator — Eurecat-Reus
Locations (1):
- Eurecat, Reus, Spain

IPD SHARING:
Plan to Share IPD: Yes
The data will be shared with other researchers involved in the MED4Youth study
Supporting Information: Study Protocol, CSR
Time Frame: Study protocol will be published in a scientific international journal. Clinical Study Report will be published at the end of the study.
Access Criteria: Data will be only shared with the researchers involved in the study. Protocol and results will be shared with scientific community

REFERENCES:
- [Background] Guideline: Assessing and Managing Children at Primary Health-Care Facilities to Prevent Overweight and Obesity in the Context of the Double Burden of Malnutrition: Updates for the Integrated Management of Childhood Illness (IMCI). Geneva: World Health Organization; 2017. Available from http://www.ncbi.nlm.nih.gov/books/NBK487902/ PMID 29578661
- [Background] Miller AL, Lee HJ, Lumeng JC. Obesity-associated biomarkers and executive function in children. Pediatr Res. 2015 Jan;77(1-2):143-7. doi: 10.1038/pr.2014.158. Epub 2014 Oct 13. PMID 25310758
- [Background] US Preventive Services Task Force; Grossman DC, Bibbins-Domingo K, Curry SJ, Barry MJ, Davidson KW, Doubeni CA, Epling JW Jr, Kemper AR, Krist AH, Kurth AE, Landefeld CS, Mangione CM, Phipps MG, Silverstein M, Simon MA, Tseng CW. Screening for Obesity in Children and Adolescents: US Preventive Services Task Force Recommendation Statement. JAMA. 2017 Jun 20;317(23):2417-2426. doi: 10.1001/jama.2017.6803. PMID 28632874
- [Background] Schroder H, Mendez MA, Ribas-Barba L, Covas MI, Serra-Majem L. Mediterranean diet and waist circumference in a representative national sample of young Spaniards. Int J Pediatr Obes. 2010 Dec;5(6):516-9. doi: 10.3109/17477161003777417. Epub 2010 Sep 23. PMID 20863166
- [Background] Velazquez-Lopez L, Santiago-Diaz G, Nava-Hernandez J, Munoz-Torres AV, Medina-Bravo P, Torres-Tamayo M. Mediterranean-style diet reduces metabolic syndrome components in obese children and adolescents with obesity. BMC Pediatr. 2014 Jul 5;14:175. doi: 10.1186/1471-2431-14-175. PMID 24997634
- [Background] Salas-Salvado J, Diaz-Lopez A, Ruiz-Canela M, Basora J, Fito M, Corella D, Serra-Majem L, Warnberg J, Romaguera D, Estruch R, Vidal J, Martinez JA, Aros F, Vazquez C, Ros E, Vioque J, Lopez-Miranda J, Bueno-Cavanillas A, Tur JA, Tinahones FJ, Martin V, Lapetra J, Pinto X, Daimiel L, Delgado-Rodriguez M, Matia P, Gomez-Gracia E, Diez-Espino J, Babio N, Castaner O, Sorli JV, Fiol M, Zulet MA, Bullo M, Goday A, Martinez-Gonzalez MA; PREDIMED-Plus investigators. Effect of a Lifestyle Intervention Program With Energy-Restricted Mediterranean Diet and Exercise on Weight Loss and Cardiovascular Risk Factors: One-Year Results of the PREDIMED-Plus Trial. Diabetes Care. 2019 May;42(5):777-788. doi: 10.2337/dc18-0836. Epub 2018 Nov 2. PMID 30389673
- [Background] Esposito K, Kastorini CM, Panagiotakos DB, Giugliano D. Mediterranean diet and weight loss: meta-analysis of randomized controlled trials. Metab Syndr Relat Disord. 2011 Feb;9(1):1-12. doi: 10.1089/met.2010.0031. Epub 2010 Oct 25. PMID 20973675
- [Background] Iaccarino Idelson P, Scalfi L, Valerio G. Adherence to the Mediterranean Diet in children and adolescents: A systematic review. Nutr Metab Cardiovasc Dis. 2017 Apr;27(4):283-299. doi: 10.1016/j.numecd.2017.01.002. Epub 2017 Jan 12. PMID 28254269
- [Background] Abbondio M, Palomba A, Tanca A, Fraumene C, Pagnozzi D, Serra M, Marongiu F, Laconi E, Uzzau S. Fecal Metaproteomic Analysis Reveals Unique Changes of the Gut Microbiome Functions After Consumption of Sourdough Carasau Bread. Front Microbiol. 2019 Jul 30;10:1733. doi: 10.3389/fmicb.2019.01733. eCollection 2019. PMID 31417524
- [Background] Stamataki NS, Yanni AE, Karathanos VT. Bread making technology influences postprandial glucose response: a review of the clinical evidence. Br J Nutr. 2017 Apr;117(7):1001-1012. doi: 10.1017/S0007114517000770. Epub 2017 May 2. PMID 28462730
- [Background] Wallace TC, Murray R, Zelman KM. The Nutritional Value and Health Benefits of Chickpeas and Hummus. Nutrients. 2016 Nov 29;8(12):766. doi: 10.3390/nu8120766. PMID 27916819
- [Background] Casas-Agustench P, Lopez-Uriarte P, Bullo M, Ros E, Cabre-Vila JJ, Salas-Salvado J. Effects of one serving of mixed nuts on serum lipids, insulin resistance and inflammatory markers in patients with the metabolic syndrome. Nutr Metab Cardiovasc Dis. 2011 Feb;21(2):126-35. doi: 10.1016/j.numecd.2009.08.005. Epub 2009 Dec 22. PMID 20031380
- [Background] Kerimi A, Nyambe-Silavwe H, Gauer JS, Tomas-Barberan FA, Williamson G. Pomegranate juice, but not an extract, confers a lower glycemic response on a high-glycemic index food: randomized, crossover, controlled trials in healthy subjects. Am J Clin Nutr. 2017 Dec;106(6):1384-1393. doi: 10.3945/ajcn.117.161968. Epub 2017 Oct 11. PMID 29021286
- [Background] Gheflati A, Mohammadi M, Ramezani-Jolfaie N, Heidari Z, Salehi-Abargouei A, Nadjarzadeh A. Does pomegranate consumption affect weight and body composition? A systematic review and meta-analysis of randomized controlled clinical trials. Phytother Res. 2019 May;33(5):1277-1288. doi: 10.1002/ptr.6322. Epub 2019 Mar 18. PMID 30882964
- [Background] Del Chierico F, Vernocchi P, Dallapiccola B, Putignani L. Mediterranean diet and health: food effects on gut microbiota and disease control. Int J Mol Sci. 2014 Jul 1;15(7):11678-99. doi: 10.3390/ijms150711678. PMID 24987952
- [Background] Hofsteenge GH, Chinapaw MJ, Delemarre-van de Waal HA, Weijs PJ. Validation of predictive equations for resting energy expenditure in obese adolescents. Am J Clin Nutr. 2010 May;91(5):1244-54. doi: 10.3945/ajcn.2009.28330. Epub 2010 Mar 17. PMID 20237141
- [Background] Castro-Quezada I, Roman-Vinas B, Serra-Majem L. The Mediterranean diet and nutritional adequacy: a review. Nutrients. 2014 Jan 3;6(1):231-48. doi: 10.3390/nu6010231. PMID 24394536
- [Background] Serra-Majem L, Ribas L, Ngo J, Ortega RM, Garcia A, Perez-Rodrigo C, Aranceta J. Food, youth and the Mediterranean diet in Spain. Development of KIDMED, Mediterranean Diet Quality Index in children and adolescents. Public Health Nutr. 2004 Oct;7(7):931-5. doi: 10.1079/phn2004556. PMID 15482620
- [Background] Ho M, Garnett SP, Baur LA, Burrows T, Stewart L, Neve M, Collins C. Impact of dietary and exercise interventions on weight change and metabolic outcomes in obese children and adolescents: a systematic review and meta-analysis of randomized trials. JAMA Pediatr. 2013 Aug 1;167(8):759-68. doi: 10.1001/jamapediatrics.2013.1453. PMID 23778747
- [Background] Kelishadi R, Gidding SS, Hashemi M, Hashemipour M, Zakerameli A, Poursafa P. Acute and long term effects of grape and pomegranate juice consumption on endothelial dysfunction in pediatric metabolic syndrome. J Res Med Sci. 2011 Mar;16(3):245-53. PMID 22091240
- [Background] Martinez-Gonzalez MA, Salas-Salvado J, Estruch R, Corella D, Fito M, Ros E; PREDIMED INVESTIGATORS. Benefits of the Mediterranean Diet: Insights From the PREDIMED Study. Prog Cardiovasc Dis. 2015 Jul-Aug;58(1):50-60. doi: 10.1016/j.pcad.2015.04.003. Epub 2015 May 1. PMID 25940230